CLINICAL TRIAL: NCT01596920
Title: A Multicenter, Adaptive Design, Randomized, Single-Blind Study With an Open-Label Extension Option to Further Evaluate the Safety and Efficacy of Grafix® for the Treatment of Chronic Diabetic Foot Ulcers
Brief Title: Grafix® DFU: Open-Label Extension Option to Evaluate Safety & Efficacy of Grafix® for Chronic Diabetic Foot Ulcers
Acronym: DFU
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Osiris Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Osiris 302
Record Dates: First submitted 2012-03-14; First posted 2012-05-11 (Estimated); Last update posted 2014-04-09 (Estimated); Status verified 2014-04

CONDITIONS: Diabetic Foot Ulcers
Keywords: Chronic DFUs; Diabetic Foot Ulcers
MeSH Terms: conditions — Diabetic Foot | interventions — Histocompatibility Testing

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Grafix® (Active Comparator)
  Interventions: Other: Tissue
- Control (non-adherent dressing) (Placebo Comparator)
  Interventions: Other: Control

INTERVENTIONS:
Other: Tissue — Allograft Tissue Cellular Repair Matrix
  Arms: Grafix®
Other: Control — Non-adherent Dressing
  Arms: Control (non-adherent dressing)

SUMMARY:
The primary objective of the present study is to further establish in a randomized controlled trial, the safety and efficacy of weekly Grafix® administration versus control in patients with chronic diabetic foot ulcers. The primary endpoint is complete wound closure of the index wound, defined as 100% re-epithelialization as determined by the Investigator.

Grafix® is a product regulated for use in the US by the FDA as a Human Cellular and Tissue Based Product (HCT/P) under Title 21 CFR Part 1271.

DETAILED DESCRIPTION:
The treatment indication is for chronic, diabetic foot ulcers (DFUs) between 1cm2 and 15cm2 located below the malleoli on the plantar or dorsal surface of the foot. Patients must have confirmed Type I or Type II Diabetes.

Patients will receive treatment every week for 12 weeks duration in the Single-Blind Treatment phase of the trial.

Patients who receive Grafix® or control will be evaluated for primary efficacy up to 84 days, and for safety and wound re-occurrence for 84 days after wound closure. Patients in the control group whose wounds are not closed at the end of treatment may be offered Grafix® in an Open-Label Treatment phase. The Open-Label Treatment phase can last up to an additional 84 days.

ELIGIBILITY:
Inclusion Criteria:

1. Between 18 years and 80 years of age inclusive, as of the date of screening
2. Confirmed diagnosis of Type I or Type II Diabetes
3. An Index Ulcer defined as chronic (presence of wound for > 4 weeks) but not present for more than 52 weeks at the Screening Visit
4. Index Ulcer is located below the malleoli on the plantar or dorsal surface of the foot
5. The Index Ulcer is between 1cm2 and 15 cm2 at the Screening Visit
6. The Index Ulcer extends into the dermis or subcutaneous tissue without evidence of exposed muscle, tendon, bone, or joint capsule
7. Wound is free of necrotic debris
8. Patient has adequate circulation to the foot as documented by either:

   * Ankle Brachial Index (ABI) > 0.70 and < 1.30, or
   * In patients with non-compressible ankle vessels defined as an ABI ≥ 1.30, a Toe Brachial Index (TBI) ≥ 0.50
   * In patients with non-compressible ankle vessels defined as an ABI ≥ 1.30 and TBI cannot be performed (e.g., toe is absent, wounds are present, or site cannot perform a TBI), a Doppler waveform in the posterior tibial or dorsalis pedis arteries at the ankle consistent with adequate flow in the foot (biphasic or triphasic) and other diagnostic confirmation of adequate flow (e.g., duplex imaging, normal pulse volume recording [PVR] testing).

Exclusion Criteria:

1. Index Ulcer is of non-diabetic pathophysiology
2. Gangrene is present on any part of the affected foot
3. Index Ulcer is over an active Charcot deformity
4. The longest dimension of the Index Ulcer exceeds 5 cm at the Baseline Visit
5. Patient is currently receiving dialysis
6. Patient has a glycated hemoglobin A1c (HbA1c) level of > 12%
7. Chronic oral steroid use > 7.5 mg daily
8. Requiring intravenous (IV) antibiotics to treat the index wound infection
9. Patient has an ulcer within 15cm of the Index Ulcer identified for study consideration
10. Patient is receiving oral or parenteral corticosteroids, immunosuppressive or cytotoxic agents
11. Patient is Human Immunodeficiency Virus (HIV) positive or has Acquired Immune Deficiency Syndrome (AIDS)
12. Current evidence of osteomyelitis, cellulitis, or other evidence of infection including fever or pus drainage from the wound site
13. Patient has active malignancy other than non-melanoma skin cancer
14. Patient's Index Ulcer has decreased by ≥ 30% during 1-week screening period as determined by criteria provided by the Wound Core Lab
15. Patient's random blood sugar is > 450 mg/dl at screening
16. Patient has untreated alcohol or substance abuse at the time of screening
17. Pregnant women
18. Patient is currently enrolled or participated in another investigational device, drug, or biological trial within 60 days of screening
19. Patient has allergy to primary or secondary dressing materials used in this trial
20. Patient has had within the last 30 days, or is currently undergoing, or is planning for wound treatments with enzymes, growth factors, living skin, dermal substitutes or other advanced biological therapies

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2012-04; Primary Completion 2013-08 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Complete closure of the index wound, defined as 100% re-epithelialization as determined by the Investigator, anytime up to the Day 84 Visit | Up to 84 days

SECONDARY OUTCOMES:
Time to initial wound closure | Up to 84 days after the Single-Blind Treatment Visits
number of patients with >50% reduction in wound size by Day 28 | Up to 84 days after the Single-Blind Treatment Visits
number of applications of Grafix® versus control | Up to 84 days after the Single-Blind Treatment Visits
number of re-occurrences of index wound post-healing | Up to 84 days after the Single-Blind Treatment Visits
percent of wounds achieving complete closure | Up to 84 days after the Single-Blind Treatment Visits

CONTACTS AND LOCATIONS:
Overall Officials: Sharron E McCulloch, Study Director — Osiris Therapeutics, Inc
Locations (15):
- United States (15):
  - Institute for Advanced Wound Care at Baptist Medical, Montgomery, Alabama
  - Clinical Trials of Arizona, Inc., Glendale, Arizona
  - ILD Laser and Research Center, Encinitas, California
  - Nature Coast Clinical Research, Inverness, Florida
  - River City Clinical Research, Jacksonville, Florida
  - Aiyan Diabetes Center, Evans, Georgia
  - Ocean County Foot and Ankle Surgical Associates, Toms River, New Jersey
  - UNC at Chapel Hill, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Ohio Health Research Institute, Columbus, Ohio
  - Blair Orthopedics Associates, Inc, Altoona, Pennsylvania
  - Omega Medical Research, Warwick, Rhode Island
  - UT Southwestern Medical Center at Dallas, Dallas, Texas
  - Clincal Trials of Texas, Inc., San Antonio, Texas